CLINICAL TRIAL: NCT03595215
Title: Posterior Tibial Nerve Stimulation's Effectiveness in UI Frequency in Overactive Patients in Home
Acronym: OAB Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD-12-1076
Record Dates: First submitted 2018-06-22; First posted 2018-07-23 (Actual); Results first posted 2020-01-03 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Overactive Bladder
Keywords: TENS
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TENS Treatment Arm (Experimental): This study is an early feasibility study which will be treating all patients at least 3 times per week, for 8 weeks, using the device.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation

SUMMARY:
This pilot clinical study, which focuses on feasibility and proof-of-principle, will be conducted in 11 female subjects (55-100 years old) with UI. Subjects will use the device three times a week for 8 weeks and complete 3-day "voiding diaries" to record instances of UI episodes and OAB quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. 55-100 years old
3. Have an average urinary frequency of ≥ 8 voids per 24 hours (based on a pre-treatment 3-day voiding "training" diary)
4. Have self-reported bladder symptoms of more than 3 months
5. Are ambulatory and able to use the toilet independently
6. Have been off antimuscarinics, anticholinergics or beta-3 agonists for at least 2 weeks prior to enrollment OR on a stable dose for the prior 3 months
7. Patient has urinary urge incontinence of ≥ 8 episodes from a 3-day diary (with incontinence associated at urge level moderate or severe)
8. Able to provide informed consent
9. Capable and willing to follow all study-related procedures

Exclusion Criteria:

1. Have primary complaint of stress urinary incontinence
2. Have a pacemaker or implantable defibrillator
3. Had botox injections in the bladder or pelvic floor muscles in the past 12 months
4. Have a current urinary tract or vaginal infection
5. Have an active implantable SNS device (InterStim & Bion)
6. Have been diagnosed with peripheral neuropathy or nerve damage
7. Currently pregnant
8. Deemed unsuitable for enrollment in study by the investigator based on subjects' history or physical examination

Ages: 55 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TENS Treatment Arm
Started | 18
Completed | 10
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | TENS Treatment Arm
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
UUI [Mean (Standard Deviation); unit: Episodes] — Urge Incontinence Episodes
  Episodes | 5.6 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urge Incontinence Episodes
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: UUI
Arm/Group | TENS Treatment Arm
Number analyzed (Participants) | 10
UUI | 3.9 (4.0)

2. Secondary Outcome: Change in Micturitions Per Day
Description: Mean number of urinary voids per day (taken over a 3-day period)
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: voids per day
Arm/Group | TENS Treatment Arm
Number analyzed (Participants) | 10
voids per day | 5.6 (13.9)

3. Secondary Outcome: Change in Health-related Quality of Life (HRQL)
Description: Change in incontinence health-related quality of life (HRQL) scores compared to pre-treatment. The survey consists of 13 questions that can be scored from 1 to 6. Lower scores correspond with better quality of life. The lowest score possible is 13 and the highest is 78.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TENS Treatment Arm
Number analyzed (Participants) | 10
units on a scale | -19.5 (14.5)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 8 weeks for each for each participant
Arm/Group | TENS Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03595215/Prot_SAP_000.pdf